CLINICAL TRIAL: NCT00266162
Title: Therapy of Pulmonary Arterial Hypertension (PAH) With Bosentan in Patients With Eisenmenger Syndrome
Brief Title: Bosentan in Treatment of Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Competence Network for Congenital Heart Defects (Other Government)
Collaborators: German Federal Ministry of Education and Research (Other Government); Actelion (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP 3.2; 01G10210
Record Dates: First submitted 2005-12-15; First posted 2005-12-16 (Estimated); Last update posted 2008-05-07 (Estimated); Status verified 2008-05

CONDITIONS: Eisenmenger Syndrome
Keywords: Heart Defects, Congenital; Eisenmenger Complex; Hypertension, Pulmonary; Pulmonary Heart Disease; Pulmonary Circulation; Vascular Resistance
MeSH Terms: conditions — Eisenmenger Complex; Heart Defects, Congenital; Hypertension, Pulmonary; Pulmonary Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bosentan administration

SUMMARY:
Eisenmenger's syndrome presents as a severe clinical picture of polymorbidity that constitutes a great burden at the individual as well as the familial and social level. The combination of critically increased pulmonary vascular resistance, progressive pressure load of the right ventricle and disturbance of pulmonary gas exchange result in long-term polymorbidity. The objective of this study is to look into the effects of medium-term pulmonary pressure-lowering treatment with oral bosentan in patients with congenital heart defects and clinically relevant pulmonary arterial hypertension (PAH), taking advantage of extensive diagnostic procedures.

DETAILED DESCRIPTION:
Eisenmenger's syndrome presents as a severe clinical picture of polymorbidity that constitutes a great burden at the individual as well as the familial and social level. The combination of critically increased pulmonary vascular resistance, progressive pressure load of the right ventricle and disturbance of pulmonary gas exchange result in long-term polymorbidity. While the patient's ability to care for him-/ herself gets lost over time, the financial burden due to the need for medical consultations and hospital stays increases. This is distressing to both the patient and the family. Usually, death results from cardiac decompensation in the presence of gradually increasing pulmonary vascular resistance and hypoxic lesion of organs including the myocardium (Hopkins, AJC 2002).

With a better understanding of the pathophysiology underlying pulmonary hypertension, novel therapeutic approaches have been developed during the past few years. These include a) inhibition of the NO-cGMP-degrading type 5 phosphodiesterase (PDE-5) and b) antagonising the endothelin system (Krum, Curr Opin Investig Drugs 2003). The goal is a dilatation of the abnormally constricted pulmonary arterial vessels by relaxation of the vascular smooth muscle cells with a reversal of pulmonary vascular remodelling (Ghofrani, Pneumologie 2002).

Specific drugs affecting pulmonary vascular resistance have been studied. Intravenous prostacyclin has major disadvantages: high cost, tachyphylaxis, risk of infection and rebound hypertension upon discontinuation. Inhalative pulmonary vasodilators, in particular iloprost, may be effective in primary pulmonary hypertension (Olschewski, Ann Int Med 1996; Hoeper, Pneumologie 2001), but administration is time-consuming, and due to its mode of application its effects are intermittent, lasting only about 75 minutes (Hoeper, JACC 2000). Considering this, oral treatments appear preferable, because of easy administration and, hence, better patient compliance.

Bosentan (Tracleer®) is a non-selective endothelin receptor antagonist with dual binding (ETA and ETB) and complete blocking of endothelin-1. It is the first drug of this class that was approved for the lowering of pulmonary vascular resistance. Significant effects on haemodynamics and exercise tolerance were demonstrated for both monotherapy (Galie, J Am Coll Cardiol 2003; Rubin, N Engl J Med 2002) and add-on treatment with inhalational and parenteral prostanoids (Hoeper, Eur Respir J 2003). In children with at least 10 kg body weight, bosentan significantly improved pulomary haemodynamics, while pharmacokinetics was found to be comparable to that in adults (Bars, Clin Pharmacol Ther 2003). Good long-term tolerability and effectiveness over a period of one year were demonstrated (Sitbon, Chest 2003). Moreover, in animal models of increased pulmonary blood flow activation of the endothelin system was absent under bosentan treatment and both haemodynamic and morphological changes were prevented. Available data suggest that the effects of bosentan are not limited to primary pulmonary hypertension. Further studies are required to prove its effectiveness in pulmonary hypertension of various aetiologies.

The objective of this study is to look into the effects of medium-term pulmonary pressure-lowering treatment with oral bosentan in patients with congenital heart defects and clinically relevant pulmonary arterial hypertension (PAH), taking advantage of extensive diagnostic procedures. The data obtained are supposed to contribute to the development of guidelines for the treatment of PAH caused by congenital heart defects. The data will be further evaluated in terms of health economics (network subproject "Health Economics", project manager: Prof. Dr. med. Karl W. Lauterbach).

The hypotheses are:

1. Bosentan specifically improves the pulomonary vascular damage caused by hypercirculation. As an immediate effect, it blocks vasoconstriction, and on the long run, it reverts pulmonary vascular remodelling.
2. In patients with Eisenmenger's syndrome, this results in a decrease in pulmonary vascular resistance and a normalization of pulmonary vascular responsiveness.
3. This is followed by an increase in lung perfusion and systemic oxygen supply.
4. The patient benefits from an improvement in his/her clinical condition and exercise tolerance.

These hypotheses will be tested by comparing findings of the following examinations before and immediately after the 24-week treatment with bosentan: clinical examination, ECG, echocardiography, CPX, MRT, cardiac catheterization with pulmonary artery manometry, and laboratory tests. As a secondary objective, the degree of concordance of findings of different invasive and non-invasive examinations and diagnostic procedures will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific:

  * Written informed consent obtained
* Specific:

  * Age at least 18 years
  * Presence of cyanosis with < 93 % arterial oxygen saturation (measured by transcutaneous pulse oximetry)
  * Clinical indication for the invasive diagnostic procedures planned for the study is given; this is evaluated on the basis of observation before, during and after medicinal treatment)
  * Presence of PAH as diagnosed by invasive methods with Rp:Rs > 0.75 measured at rest, before testing of pulmonary vasodilatory reserve
  * One of the following diagnoses:

    * non-corrected large congenital shunting defect at atrial, ventricular or arterial level: PAPVD, ASD, SVD, VSD, AVSD, TAC, APW, PDA, or a combination of these.
    * Surgically corrected shunting defect (diagnoses as above) with significant residual defect
    * Other diagnoses with univentricular physiology/haemodynamics.

Exclusion Criteria:

* Non-specific:

  * pregnancy or lactation
  * women of child-bearing age who are sexually active without practising reliable methods of contraception
  * any disease or impairment that, in the opinion of the investigator, excludes a subject from participation
  * substance abuse (alcohol, medicines, drugs)
  * other medical, psychological or social circumstances that would adversely affect a patient's ability to participate adequately in the study or increase the risk to the patient or others in the case of participation.
  * insufficient compliance
  * subjects in whom MRI cannot be performed (contrast medium allergy, claustrophobia, cardiac pacemaker)
  * subjects who are not able to perform CPX
* Specific:

  * pulmonary hypertension of any aetiology other than those specified in the inclusion criteria
  * subjects with known intolerance of NO or iloprost or their constituents
  * acute decompensated heart failure within 7 days before the invasive procedure
  * haemodynamic instability that would increase the risk of pulmonary arterial reactivity testing
  * arterial hypotension
  * anaemia (Hb < 10 g/dl)
  * decompensated symptomatic polycythaemia
  * thrombocytopenia (< 50,000/μl)
  * secondary impairment of organic (renal, hepatic) function
  * other sources of pulmonary blood flow which render the measurement of the blood flow to the lungs and pulmonary vascular resistance impossible
  * obstruction of pulmonary blood outflow
  * left ventricular diseases
  * significant valvular diseases other than tricuspid or pulmonary regurgitation
  * pericardial constriction
  * history of stroke, myocardial infarction or life-threatening arrhythmia within 6 months before screening
  * bronchopulmonary dysplasia or other chronic lung diseases
  * history of significant pulmonary embolism
  * other relevant diseases (e.g. HIV infection)
  * trisomy 21
  * Prohibited concomitant medication: Any medication listed below which has not been discontinued at least 30 days prior to screening.
  * Unspecified or other significant medication (e.g. medication for diabetes or immunosuppression)
  * Unstable medication, recent changes in dosage regimen
  * Drugs to treat pulmonary hypertension (endothelin receptor antagonists, PDE-5 antagonists, prostanoids. (Specific pulmonary vasodilators during cardiac catheterisation are allowed.)
  * Other medication with vascular action
  * Medication that is not compatible with bosentan or that interferes with its metabolism (inhibitors of CYP2C9 or CYP3A4) or that, in the investigator's opinion, may interfere with bosentan treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2004-08; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
maximal exercise tolerance (walking distance in the 6-minute walking test)
peripheral oxygen saturation (SatO2)
pulmonary-systemic ratio of arterial resistance (Rp:Rs)

SECONDARY OUTCOMES:
NYHA class
increase in pulmonary reagibility by bosentan therapy
normalisation of vasoactive mediators by bosentan therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ingram Schulze-Neick, MD, Principal Investigator — German Heart Institute
Locations (8):
- Germany (8):
  - Kinderkardiologie Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - Universitätsklinikum Giessen and Marburg, Giessen, Hesse
  - Herz-und Diabeteszentrum NRW, Bad Oeynhausen, North Rhine-Westphalia
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel, North Rhine-Westphalia
  - Universitätsklinikum des Saarlandes, Homburg, Saarland
  - Universitätsklinikum der Martin-Luther-Universität Halle-Wittenberg, Halle, Saxony-Anhalt
  - Deutsches Herzzentrum Berlin, Berlin, State of Berlin